CLINICAL TRIAL: NCT04674072
Title: The Effect of the Reverse Nordic Curl Exercise on Quadriceps Femoris Muscles Injuries Rate Among Soccer Players: Cluster Randomized Controlled
Brief Title: The Effect of the Reverse Nordic Curl Exercise on Quadriceps Femoris Muscles Injury Rate Among Soccer Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Wesam Saleh A. Al Attar, PT, MSc, PhD, Professor, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HAPO-02-K-012-2020-11-480
Record Dates: First submitted 2020-12-08; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Quadriceps Tendon Rupture; Quadriceps Strained Tendon; Quadriceps Muscle Atrophy
Keywords: Injury Prevention Program; Reverse Nordic curl exercise

STUDY DESIGN:
Intervention Model Description: The intervention group will be instructed to include the reverse Nordic curl exercise into their warm up 15 to 20 mins before training session (3 times per week) during one season (6 months).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will be instructed to include the reverse Nordic curl exercise into their warm up 15 to 20 mins before training session (3 times per week) during one season (6 months).
  Interventions: Other: Reverse Nordic curl exercise
- Control group (Active Comparator): The control group will practice their usual warm up. Usual warm up is defined as any basic exercises performed before a performance or practice to prepare the muscles for vigorous actions
  Interventions: Other: Usual warm up

INTERVENTIONS:
Other: Reverse Nordic curl exercise — The reverse Nordic curl is a body-weight exercise which mainly works the quadriceps and hip flexors. It has a large eccentric component, meaning the muscles are working whilst lengthening.
  Arms: Intervention group
Other: Usual warm up — Usual warm up is defined as any basic exercises performed before a performance or practice to prepare the muscles for vigorous actions.
  Arms: Control group

SUMMARY:
The reverse Nordic curl is a body-weight exercise which mainly works the quadriceps and hip flexors. It has a large eccentric component, meaning the muscles are working whilst lengthening.

The purpose of this study is to investigate the effect of the reverse Nordic curl exercise on Quadriceps femoris muscles injuries among soccer players.

It hypothesized that reverse Nordic curl exercise has a beneficial effect in terms of Quadriceps femoris muscles injury prevention.

DETAILED DESCRIPTION:
Description of intervention(s) / exposure The intervention group will be instructed to include the reverse Nordic curl exercise into their warm up 15 to 20 mins before training session (3 times per week) during one season (6 months).

Group sessions will be administered by an exercise physiologist and/ or athletic trainer and/ or soccer coaches and/ or strength and conditioning specialists and/ or physiotherapist.

Session attendance checklists will be used to assess or monitor adherence to the intervention.

The reverse Nordic curl is a body-weight exercise which mainly works the quadriceps and hip flexors. It has a large eccentric component, meaning the muscles are working whilst lengthening.

This is a very simple movement to do, but maintaining strict positioning is vital to get the full benefits. Here's how to do it:

Grab a mat on a soft floor. Kneel down, and sit on top of the feet. If trying this exercise for the first time, place the knees and feet close together, approximately hip-width apart. For more advanced, the feet and knees slightly wider, just outside the hips, to be able to lay back farther without hitting the legs.

Sit up in a tall kneeling position, push the hips forward, and lock the rib cage down. Looking to create a straight line down the front of the body, especially at the hips. This is to create a stretch at the hip flexor muscles.

Lower the shoulders towards the floor by bending at the knee, maintaining the "plank" position previously created. If hip extension is maintained, and the core adequately braced, there should be no strain on the low back, and an intense stretch felt down the front of the legs.

Continue to lean back as far as it is possible to control, then squeeze the quads to return to the starting position (this may not be very far to begin with). It is crucial to NOT let the hips drop backwards at any point during the movement. If they do, the stretch on the hip flexors will be released, defeating the point of the exercise.

Once reaching the floor and back is possible for multiple sets of 10+ repetitions, can begin loading the movement by holding a light plate, kettlebell or dumbbell.

ELIGIBILITY:
Inclusion Criteria:

* Soccer teams
* Amateur.
* Male .
* Training at least three times per week.

Exclusion Criteria:

* History of lower extremity injury requiring medical attention in the past 6 months, or systemic diseases, cardiovascular disease, neurological disorders or bone fractures or surgery in the previous year.

Players who joined a participating team after the start of the trial will be excluded.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-01-16 (Estimated); Primary Completion 2021-06-16 (Estimated); Study Completion 2021-07-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of initial injuries | At the end of the intervention season (6 months).
  Injury is defined according to a consensus statement on injury definitions and data collection procedures in soccer studies; an injury will be recorded if it caused the player to be unable to completely participate in the following match or training session.
  Coaches in both the experimental and control groups will be reporting injuries during training and matches by filling in forms once per week and submitting the information using the Sports Injury Tracker injury reporting form (Sports Medicine Australia).
  Injury rates will be summarised as number of injuries per 1000 player-hours for both matches and training. Exposure time in hours will be calculated for each team over a 6-month period.
The incidence of recurrent injuries | At the end of the intervention season (6 months)
  Recurrent injury is defined as a repeat episode of a fully recovered injury. Injury is defined according to a consensus statement on injury definitions and data collection procedures in soccer studies; an injury will be recorded if it caused the player to be unable to completely participate in the following match or training session.
  Coaches in both the experimental and control groups will be reporting injuries during training and matches by filling in forms once per week and submitting the information using the Sports Injury Tracker injury reporting form (Sports Medicine Australia).
  Injury rates will be summarised as number of injuries per 1000 player-hours for both matches and training. Exposure time in hours will be calculated for each team over a 6-month period.

SECONDARY OUTCOMES:
Injury severity | At the end of the intervention season (6 months)
  Defined as time loss in days (days unable to train): minor (1 to 7 days lost), moderate (8 to 21 days lost), or severe (>21 days lost). Injury severity data will be collected from Sports Injury Tracker injury reporting form.
Compliance with the intervention | At the end of the intervention season (6 months)
  The rate of compliance using attendance log

CONTACTS AND LOCATIONS:
Locations (1):
- Umm Al Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Start: Immediately following publication. End: No end date determined.
Access Criteria: Access subject to approvals by Principal Investigator. The Principal Investigator can be contacted by email wsattar@uqu.edu.sa

REFERENCES:
- [Background] Alonso-Fernandez D, Docampo-Blanco P, Martinez-Fernandez J. Changes in muscle architecture of biceps femoris induced by eccentric strength training with nordic hamstring exercise. Scand J Med Sci Sports. 2018 Jan;28(1):88-94. doi: 10.1111/sms.12877. Epub 2017 Apr 10. PMID 28314091
- [Result] Al Attar WSA, Soomro N, Sinclair PJ, Pappas E, Sanders RH. Effect of Injury Prevention Programs that Include the Nordic Hamstring Exercise on Hamstring Injury Rates in Soccer Players: A Systematic Review and Meta-Analysis. Sports Med. 2017 May;47(5):907-916. doi: 10.1007/s40279-016-0638-2. PMID 27752982